CLINICAL TRIAL: NCT02104479
Title: Open Multicenter Diagnostic Study on the Accuracy of Biomarker Testing (Galactomannan (GM), (1-3)-β-D-glucan (BDG), Aspergillus-specific Polymerase Chain Reaction (PCR) Assay) in Pleural Effusion Samples of Immunocompromised Patients With Suspected Invasive Pulmonary Aspergillosis (IPA)
Brief Title: Diagnostic Accuracy of Pleural Effusion Aspergillosis Biomarker Testing
Acronym: EFFU-ASP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Heidelberg University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dieter Buchheidt, MD, Heidelberg University
Other Study IDs: EFFU-ASP 2014
Record Dates: First submitted 2014-03-27; First posted 2014-04-04 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Invasive Aspergillosis; Pleural Effusion; Immunosuppression
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — only fungal DNA is investigated, no human DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Immunocompromised Patients: Immunocompromised patients with suspected IPA who have Pleural effusions act as the observed study population
- Control Group: Patients without Immunosuppression with pleural effusions

SUMMARY:
Diagnostic accuracy of biomarker testing (galactomannan (GM), (1

DETAILED DESCRIPTION:
A multicentre, open, prospective diagnostic study on the diagnostic accuracy of biomarker testing (galactomannan (GM), (1

ELIGIBILITY:
Inclusion Criteria:

* prolonged neutropenia > 10 d, patients
* after allogeneic stem cell transplantation or solid organ transplantation,
* Patients wth acute leukemia in induction treatment,
* patients witrh graft-versus-host-disease,
* patients under chronic immunusuppressive therapy such as ciclosporin,
* patients with HIV,
* patients with chronic steroid treatment

Exclusion Criteria:

* Age < 18 years
* missing informed consent
* contraindication for pleural centesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Immunocompomised Patients based on the following conditions: prolonged neutropenia > 10 d, patients after allogeneic stem cell transplantation or solid organ transplantation, Patients wth acute leukemia in induction treatment, patients witrh graft-versus-host-disease, patients under chronic immunusuppressive therapy such as ciclosporin, patients with HIV, patients with chronic steroid treatment,
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-03-31 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Test Sensitivity | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Buchheidt, MD, Principal Investigator — Universitätsmedizin Mannheim
Locations (2):
- Germany (2):
  - University Hospital Mannheim, Mannheim, Baden-Wuerrtemberg
  - Wuerzburg University Hospital, Würzburg, Bavaria

REFERENCES:
- [Background] Reinwald M, Spiess B, Heinz WJ, Heussel CP, Bertz H, Cornely OA, Hahn J, Lehrnbecher T, Kiehl M, Laws HJ, Wolf HH, Schwerdtfeger R, Schultheis B, Burchardt A, Klein M, Durken M, Claus B, Schlegel F, Hummel M, Hofmann WK, Buchheidt D. Aspergillus PCR-based investigation of fresh tissue and effusion samples in patients with suspected invasive Aspergillosis enhances diagnostic capabilities. J Clin Microbiol. 2013 Dec;51(12):4178-85. doi: 10.1128/JCM.02387-13. Epub 2013 Oct 9. PMID 24108612